CLINICAL TRIAL: NCT01868087
Title: Impact Advanced Recovery® for Radical Cystectomy (RC) Patients
Brief Title: Impact Advanced Recovery® for Radical Cystectomy (RC) Patients: a Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jill Hamilton-Reeves, PhD RD LD (Other)
Collaborators: American Cancer Society, Inc. (Other); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor-Investigator, Jill Hamilton-Reeves, PhD RD LD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13730
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer; Radical Cystectomy; Urinary Bladder Neoplasms; Surgery
Keywords: nutritional supplement; immune system; RC surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impact Advanced Recovery® (Experimental): 3 briks daily (240 mL per brik) of Impact Advanced Recovery® to be take for 5 days before and after RC surgery
  Interventions: Dietary Supplement: Impact Advanced Recovery®
- Boost Plus® (Placebo Comparator): 3 briks daily (240 mL per brik) of Boost Plus® to be take for 5 days before and after RC surgery
  Interventions: Dietary Supplement: Boost Plus®

INTERVENTIONS:
Dietary Supplement: Boost Plus®
  Arms: Boost Plus®
Dietary Supplement: Impact Advanced Recovery®
  Arms: Impact Advanced Recovery®

SUMMARY:
The purpose of this study is determine if using Impact Advanced Recovery® before and after RC surgery helps reduce surgical complications.

DETAILED DESCRIPTION:
Radical cystectomy (RC) is the removal of the entire bladder and nearby organs that may contain cancer cells. It is a major surgery that can lead to breakdown of proteins in the body and a decreased immune response, both of which increase the risk of illness and death. Poor nutrition status before RC surgery is linked to a higher rate of death after surgery. Therefore, it is important to eat a balanced diet before and after RC surgery to avoid negative outcomes.

Studies show that patients who drink a nutritional supplement that may enhance the immune system before and after gastro-intestinal surgery may have fewer infections and shorter hospital stays after surgery. Patients with cancer of the colon/rectum, stomach, and pancreas who drank a similar immune-enhancing nutritional supplement before and after surgery also had fewer infections.

The purpose of this study is to attain pilot data for a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing RC surgery for primary bladder cancer

Exclusion Criteria:

* Patients with swallowing difficulties or unable to tolerate oral intake
* Evidence of metastatic disease
* Weight loss ≥ 10% (with respect to usual body weight) in the 6 months prior to surgery or BMI ≤ 18.5
* Patients undergoing cystectomy for non-bladder primary malignancy or cancer type other than urothelial
* Active viral infections such as Human immunodeficiency virus (HIV) positive, hepatitis, or who have a known immunodeficient state
* Prior history of gouty arthritis or uric acid stones
* Patients with milk, soy, or fish allergies

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Immune and Inflammation Response | Change from Baseline to Day 30
  Measure ability of Impact Advanced Recovery® to alter body's immune and inflammation response.

SECONDARY OUTCOMES:
preservation of body weight and fat free mass (FFM) | Change from Baseline to 30 Days
  measure of body weight and fat free mass between groups over course of the study
count of infections after surgery | Change from Baseline to 30 Days
  count of total number of infections affecting study participants
hospital readmission rate | Change from Baseline to 30 Days
  readmissions required for study partipants

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton-Reeves, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Hamilton-Reeves JM, Bechtel MD, Hand LK, Schleper A, Yankee TM, Chalise P, Lee EK, Mirza M, Wyre H, Griffin J, Holzbeierlein JM. Effects of Immunonutrition for Cystectomy on Immune Response and Infection Rates: A Pilot Randomized Controlled Clinical Trial. Eur Urol. 2016 Mar;69(3):389-92. doi: 10.1016/j.eururo.2015.11.019. Epub 2015 Nov 30. PMID 26654125